CLINICAL TRIAL: NCT03640650
Title: Economic Impact of Dropless Therapy Versus Usual Care for Cataract Surgery: A Real-World Study.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID-19 pandemic leading to uncertainty in the recruitement
Sponsor: PeriPharm (Other)
Collaborators: Advance Dosage Forms, Inc. (Industry); Imprimis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PRE1701
Record Dates: First submitted 2018-05-10; First posted 2018-08-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Cataract Surgery
Keywords: Sequential bilateral cataract surgery
MeSH Terms: interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dropless Therapy (Experimental): Single used, pre-mixed, centrally compounded injectable that contains 15 mg/ml of triamcinolone acetonide and 1 mg/ml of moxifloxacin. This preservative-free suspension is injected at a dose of 0.2 mg into the posterior chamber, for a total drug delivery of 3 mg of triamcinolone acetonide and 0.2 mg of moxifloxacin. At the time of cataract surgery, Dropless is intended to be injected as a single administration into the anterior vitreous after the insertion of the IOL implant, with a 27 or 30-gauge cannula via a transzonular or transsceral pars plana injection, just before rinsing the viscoelastic fluid.
  Interventions: Combination Product: Dropless Therapy
- Usual Care (Active Comparator): This therapy usually comprises an antibiotic, a steroid and in some cases a nonsteroidal anti-inflammatory drug (NSAID). Antibacterial drops are usually given at the end of surgery and are continued for one week after the surgery. Steroid drops are usually started the day of surgery and then tapered down over 3 to 4 weeks. When prescribed, NSAIDs are usually started 2 or 3 days before surgery, or started the day of surgery, and continued for 3 or 4 times a day for 3 to 4 weeks.
  Interventions: Drug: Usual Care

INTERVENTIONS:
Combination Product: Dropless Therapy — The Dropless will be injected, as a single administration, into the vitreous cavity during the cataract surgery.
  Other Names: Triamcinolone acetonide (15mg/ml); Moxifloxacine (1mg/ml)
  Arms: Dropless Therapy
Drug: Usual Care — In order to reflect real-world clinical practice, the choice of topical ophthalmic medications as well as dosage, posology, and duration of treatment will be left to the discretion of the treating ophthalmologist.
  Other Names: Antibacterial eye drops; Nonsteroidal anti-inflammatory eye drops; Steroid eye drops
  Arms: Usual Care

SUMMARY:
This real-life Health Economics and Outcome Research (HEOR) study will enable to evaluate the economic impact of Dropless therapy for the prophylactic treatment of inflammation and infection after routine cataract surgery. This prospective randomized controlled crossover open-label study will estimate resource utilization and cost attributable to patients' management following a cataract surgery and until last follow-up visit and adherence, satisfaction and preference between usual care and Dropless in a real-life setting.

Data collected will include patients' characteristics and demographics, medical information, cataract surgery information, healthcare resource utilization, patients' adherence to topical ophthalmic medications as well as patients' satisfaction to both treatment and preference between usual care and Dropless. Patients will fill a set of questionnaires at their recruitment in the study and at their last follow-up visit for their two cataracts surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. Undergoing delayed sequential bilateral cataract extraction with intraocular lens implantation;
3. Delayed sequential bilateral cataract surgery performed in a day surgery setting;
4. Second cataract surgery planned within 3 months following the date of the first cataract surgery;
5. Ability to read and understand English or French;
6. Signature of ICF.

Exclusion Criteria:

1. Patients with other ophthalmic conditions such as glaucoma, corneal disease, agerelated macular degeneration, and active uveitis* (*In line with current clinical practice in Canada, uveitis should be inactive for 3 months to be included in the study);
2. Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation;
3. Participation in any investigational ophthalmic-related drug or device trial within the 30 days prior to the start date of this trial or participation in any current investigational ophthalmic-related drug or device trial;
4. Patients with any history of allergy to the usual care post-operative eye drops or the components of Dropless.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Cataract surgery - related healthcare resource use assessed by number of relevant medications | 30 to 45 days following each cataract surgeries
  Chart abstracted and self-reported by participant
Cataract surgery - related healthcare resource use assessed by number of medical visits (outpatient and inpatient visits) | 30 to 45 days following each cataract surgeries
  Chart abstracted and self-reported by participant
Cataract surgery - related healthcare resource use assessed by number of hospitalizations (ICU and non-ICU) | 30 to 45 days following each cataract surgeries
  Chart abstracted and self-reported by participant
Cataract surgery - related health care resource use assessed by lengths of hospital stay (ICU and non-ICU) | 30 to 45 days following each cataract surgeries
  Chart abstracted and self-reported by participant
Cataract surgery - related health care resource use assessed by number of emergency department visit | 30 to 45 days following each cataract surgeries
  Chart abstracted and self-reported by participant
Cataract surgeries - related health care resource use assessed by number of home visit from nurse | 30 to 45 days following each cataract surgeries
  Chart abstracted and self-reported by participant

SECONDARY OUTCOMES:
Medication adherence | 30 to 45 days following each cataract surgeries
  The investigator will question the participant on his adherence to drop regimen. Descriptive results of the adherence, based on self-reported adherence, will be reported in accordance to patients' responses for each question.
Medication satisfaction | 30 to 45 days following each cataract surgeries
  The investigator will question the patient in order to describe the satisfaction to drop regimen or Dropless. Descriptive results of the satisfaction, based on self-reported satisfaction, will be reported in accordance to patients' responses for each question.
Medication preference | Through study completion, an average of 20 weeks for each patient
  The investigator will question the patient about his preference between the usual care (eye drops) and Dropless. Descriptive results of the preference will be reported in accordance to patients' responses.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - CIUSSS de l'Est-de-l'Île-de-Montréal (Hôpital Maisonneuve-Rosemont), Montreal, Quebec
  - McGill Academic Eye Center, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No